CLINICAL TRIAL: NCT00160095
Title: Patient Selection for Hypoxia Modifying Treatments Based on Functional Microregional Imaging of Tumor Vasculature, Oxygenation and Proliferation in Squamous Cell Carcinoma of the Larynx
Brief Title: Patient Selection for Hypoxia Modifying Treatments in Larynx Carcinomas
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: 088; KUN 2003-2899
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Larynx Cancer
Keywords: larynx carcinoma; Tumor hypoxia; microregional imaging; hypoxia modifying treatment
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor biopsies

SUMMARY:
The purpose of this study is to identify in a prospective manner microregional profiles of oxygenation and proliferation based on exogenous and endogenous markers that are predictive for outcome of radiotherapy in squamous cell carcinoma of the larynx and to investigate if these profiles can identify patients that are most likely to benefit from hypoxia modifying treatment strategies like ARCON (Accelerated radiotherapy combined with carbogen breathing and nicotinamide).

DETAILED DESCRIPTION:
Purpose

Prognostic indicators discriminate patients with good and bad prognosis. Predictive assays are tools that select patients for specific treatments or treatment modifications such that outcome will be improved relative to conventional treatment. In oncology, many prognostic indicators based on clinical or biological tumor characteristics have been described but only very few have proven to be useful as predictive assays. We have developed an imaging modality for coregistration of tumor oxygenation and proliferation at the microregional level with preservation of the tumor anatomy and the microenvironmental structure. We have strong indications that this functional imaging can be a powerful tool for identifying those patients that will profit from hypoxia modifying treatments.

Tumor oxygenation and proliferation are recognized as important determinants of the outcome of radiotherapy and possibly also of other treatment modalities in a number of tumor types and in particular in squamous cell carcinomas. Various exogenous and endogenous markers for hypoxia and proliferation are currently available which can be studied in relation to each other, the tumor architecture and the tumor microenvironment using immunohistochemistry and advanced image analysis techniques.

The purpose of this project is to identify microregional profiles of oxygenation and proliferation based on exogenous and endogenous markers that:

1. Are predictive for outcome of radiotherapy in squamous cell carcinoma of the larynx.
2. Can identify the patients that are most likely to benefit from hypoxia modifying treatment strategies.

   And to:
3. Validate these marker profiles in a prospective manner and in a sufficiently large group of patients.

Plan of investigation

In 2001 a multicenter randomized trial was initiated comparing accelerated radiotherapy with carbogen and nicotinamide as hypoxic modifiers against accelerated radiotherapy alone in patients with carcinoma of the larynx. This trial is approved and supported by the Dutch Cancer Society and currently 6 Dutch and 1 British center are participating. This trial provides a unique opportunity to prospectively test oxygenation and proliferation related marker profiles in a large homogeneous patient population and to assess the predictive capacity in a comparative setting with one group of patients receiving a hypoxia modifying treatment and the other group not.

Paraffin-embedded biopsy specimens will be collected from all patients entered in this trial. In part of the patients, biopsies will be taken after injection of the hypoxic marker pimonidazole and the S-phase marker iododeoxyuridine (IdUrd). Sections will be immunohistochemically processed and stained for various combinations of vascular markers, endogenous hypoxia and proliferation markers and, if applicable, for pimonidazole and IdUrd. The sections will be analyzed by computerized image processing. Apart from overall single parameter values that will be obtained, the interrelationship of the various parameters will be studied and the microregional phenotype of the tumors will be characterized by quantification and integration of the marker profiles. The information thus obtained will be related to treatment outcome in terms of both local control and survival and results from the two treatment groups will be compared.

Possible results

This investigation can identify oxygenation and proliferation related parameters and profiles that are predictive for outcome of radiotherapy in squamous cell carcinoma of the larynx and provide a selection tool for hypoxia modifying treatments. The principle of characterization of the tumor phenotype at the microregional level using functional imaging may also be applied to other tumor types and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmed squamous cell carcinoma of the larynx.
* TNM-classification (UICC 1997, appendix I):
* T3-4 glottic or supraglottic carcinoma
* T2 glottic carcinoma with impaired cord mobility or subglottic extension
* T2 supraglottic carcinoma with invasion of mucosa of base of tongue or vallecula or invasion of the medial wall of the piriform sinus.
* any N-stage, M0.
* WHO performance status 0 or 1.
* Age > 18 years.
* Written informed consent.
* Treatment in the ARCON phase III trial

Exclusion Criteria:

* Prior or concurrent treatment for this tumour.
* Severe stridor and adequate debulking of airway not possible.
* Impaired renal function: serum creatinine above upper normal limit.
* Use of nephrotoxic medication (including ACE-inhibitors) that cannot be discontinued for the duration of the radiation treatment.
* Impaired hepatic function: ASAT and ALAT more than 1.5 times the upper normal limit.
* Use of anti-convulsants that cannot be discontinued for the duration of the radiation treatment.
* History of malignancy during the previous 5 years except basal cell carcinoma of skin, carcinoma in situ of the cervix, or superficial bladder neoplasm (pTa).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Squamous cell carcinoma of the larynx
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2001-07; Primary Completion 2010-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes HA Kaanders, M.D., Ph.D., Principal Investigator — Radboud University Nijmegen Medical Centre, Dept Radiation Oncology
Locations (5):
- Netherlands (5):
  - Free University Medical Centre Amsterdam, Amsterdam
  - Rijnstate Ziekenhuis Arnhem, Arnhem
  - Academic Hospital Maastricht, Maastricht
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Universitair Medisch Centrum Utrecht, Utrecht